CLINICAL TRIAL: NCT01186874
Title: Epidemiology Research on Acute Lung Injury/Acute Respiratory Distress Syndrome (ALI/ARDS) in Adult ICU in Shanghai
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Zhang Xiangyu, Director, professor, Tongji University
Other Study IDs: OARSIS20100808
Record Dates: First submitted 2010-08-09; First posted 2010-08-23 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2010-07

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To survey the prevalence and the mortality of the Acute Lung Injury/ Acute Respiratory Distress Syndrome (ALI/ARDS) in 12 university hospital ICUs in Shanghai.

DETAILED DESCRIPTION:
Acute lung injury is a critical illness syndrome consisted of acute hypoxemic respiratory failure with bilateral pulmonary infiltrates that are not attributed to left atrial hypertension. The severity of the hypoxemia differentiates these two entities, with a ratio of partial pressure of oxygen in arterial blood (PaO2) to inspired fraction of oxygen (FIO2) of less than 200 mm Hg for ARDS and of less than 300 mm Hg for ALI.[1] Although ARDS initially was reported in 1967 by Ashbaugh and colleagues[2], it was not until 1992 that the American-European Consensus Conference (AECC) on ARDS developed a standardized definition for ARDS and ALI. There are many epidemiologic researches about the incidence and mortality of the ALI/ARDS.[3-6] Gorden D [3] reported that a total of 1113 King County residents undergoing mechanical ventilation met the criteria for acute lung injury and were 15 years of age or older. On the basis of this figure, the crude incidence of acute lung injury was 78.9 per 100,000 person-years and the age-adjusted incidence was 86.2 per 100,000 person-years. The in-hospital mortality rate was 38.5 percent. In our country, Yueming Lu [7] reported in-hospital and 90-day mortalities of ARDS patients were 68.5 and 70.4% in Shanghai ICU in 2004.

In recent years, significant progress has been made in the diagnosis and treatment of the ALI/ARDS, such as the application of the lung protective ventilation strategy and the CRRT, which may prove the symptoms and the prognosis of the ALI/ARDS. However, controversies still remained. Ventilation drive pressure, early application of neuromuscular blockade, strategy of PEEP level are frequently met questions in routine practice. In our country, a guideline for the treatment and diagnosis of ALI/ARDS was developed in 2006 [8]. So the incidence and the mortality of this disease are unknown in our country now. Therefore, the investigators will perform a prospective, multi-center study to survey the incidence, risk factors and outcome of ALI/ARDS in 13 adult ICU in Shanghai.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with ALI/ARDS who are admitted to the study ICUs between 1st Aug. 2010 at 00:00 hours (midnight) and the finish date of 31st Jan. 2011 at 23:59 hours (11.59 pm). Patients who are already in the ICUs prior to 1st Aug. 2010 at 00:00 hours will not be included in the study.

Exclusion Criteria:

* Patients less than 15 years old.
* Patients with the organ transplantation, end-stage of the malignant tumors and brain death.
* The GCS of the patient is less than 8.
* Patients with severe sepsis who were directly transferred to the study ICUs from another hospital or another ICU.
* For all patients who are discharged from the ICU and readmitted to the ICU again during the study period, only the first admission during the study period will be included.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients with ALI/ARDS who are admitted to the study ICUs
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xiangyu Zhang, MD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China